CLINICAL TRIAL: NCT01097889
Title: Evaluating the Relative Effectiveness of Two Feeding Interventions for the Treatment of Moderate Acute Malnutrition in Children 6-60 Months of Age in Southern Ethiopia
Brief Title: Evaluating the Relative Effectiveness of Two Feeding Interventions for the Treatment of Moderate Acute Malnutrition
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The Hospital for Sick Children (Other)
Responsible Party: Principal Investigator, Stanley Zlotkin, Chief, Global Child Health, The Hospital for Sick Children
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 1000013545
Record Dates: First submitted 2010-03-31; First posted 2010-04-02 (Estimated); Last update posted 2021-04-19 (Actual); Status verified 2021-04

CONDITIONS: Child Nutrition Disorders
Keywords: United Nations World Food Programme; blended food (CSB); ready-to-use supplementary foods (RUSF); Plumpy®
MeSH Terms: conditions — Child Nutrition Disorders | interventions — Placental Lactogen

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Treatment Group 1 (Active Comparator)
  Interventions: Dietary Supplement: Fortified blended foods, Corn Soya Bean Flour (CSB) with oil.
- Treatment Group 2 (Experimental)
  Interventions: Dietary Supplement: RUSF (ready-to-use supplementary foods) Supplementary Plumpy®

INTERVENTIONS:
Dietary Supplement: Fortified blended foods, Corn Soya Bean Flour (CSB) with oil. — A daily ration equivalent of 300g CSB and 32g vegetable oil Bi-weekly distribution of premix of 4.2kg CSB with 0.5L vegetable oil. Estimated 1413 kcal, 47g protein
  Arms: Treatment Group 1
Dietary Supplement: RUSF (ready-to-use supplementary foods) Supplementary Plumpy® — Peanut-based fortified supplement
  One 92g sachet eaten throughout the day Bi-weekly distributions of 14 sachets 500 kcal and 13g protein
  Arms: Treatment Group 2

SUMMARY:
Supplementary feeding programs for children with moderate acute malnutrition have been implemented in developing countries using treatment foods with minimal or no evidence of their effectiveness. Fortified peanut paste is a popular new treatment food for children with severe and moderate malnutrition.

Objectives: To investigate the relative effectiveness of two non-identical therapeutic foods in children with moderate malnutrition by comparing differences in performance indicators (i.e. recovery rates), recovery times, and change in weight-for-height z-scores in each group.

This proposed research project will evaluate the relative effectiveness of two non-identical treatment foods for the treatment of moderate acute malnutrition in children

DETAILED DESCRIPTION:
This research protocol will be embedded as a component of the UN World Food Programme (WFP) -supported Supplementary Feeding programmes in Ethiopia. The proposed study is a prospective cluster-randomized equivalence trial that will compare the relative effectiveness of two feeding interventions in four woredas (districts). Research will be implemented in two comparable woredas (one with CSB and one with RUSF), in two different areas in Sidama zone that represent different livelihood zones, main source of crop income, and level of food insecurity

ELIGIBILITY:
Inclusion Criteria:

* All children 6 to 60 months of age who are identified as malnourished based on MUAC measurements with WFH ≥70 to <80%.

Exclusion Criteria:

* Children with WFH < 70% or presenting with bilateral pitting oedema (they will be referred to therapeutic feeding programme).
* Children with any illness or clinical condition that prevents them from safely ingesting either supplementary foods. A child is medically assessed upon admission for any complicated clinical condition (oedema, malaria, vomiting, chronic diarrhea, infections, appetite, etc) that would require medical care and those children will be referred to the therapeutic feeding programme.
* All children transferred from the therapeutic feeding programme directly into the supplementary feeding programme - however they will not be included in the research study.
* Children with WFH > 80% but MUAC 110 to 120 mm- they will be admitted to SFP however will not be included in the research study.

Ages: 6 Months to 60 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 2600 (Actual)
Dates: Start 2009-04 (Actual); Primary Completion 2009-11 (Actual); Study Completion 2010-07 (Actual)

PRIMARY OUTCOMES:
Survival Analysis | Baseline and at 16 Weeks
  Recovery rates in children from malnutrition

SECONDARY OUTCOMES:
Anthropometrics Changes | Baseline, Weeks 2,4,6,8,10,12,14,16
  Height, weight and middle upper arm circumference (MUAC)
Household Practices Questionnaire | At 16 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Stanley Zlotkin, MD, Principal Investigator — The Hospital for Sick Children
Locations (2):
- The Hospital for Sick Children, Toronto, Ontario, Canada
- Regional Health Board - Health Posts in South Nations and Nationalities Peoples Region (SNNPR, Sidama Zone, Southern Ethiopia, Ethiopia

REFERENCES:
- [Derived] Karakochuk C, van den Briel T, Stephens D, Zlotkin S. Treatment of moderate acute malnutrition with ready-to-use supplementary food results in higher overall recovery rates compared with a corn-soya blend in children in southern Ethiopia: an operations research trial. Am J Clin Nutr. 2012 Oct;96(4):911-6. doi: 10.3945/ajcn.111.029744. Epub 2012 Sep 5. PMID 22952175